CLINICAL TRIAL: NCT06485154
Title: Post-Injectable Cabotegravir Antiretroviral Salvage Strategy Options Trial
Acronym: PICASSO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Professor Francois Venter, Executive Director: Ezintsha, University of Witwatersrand, South Africa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EZ-BB-036
Record Dates: First submitted 2024-06-10; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: HIV Prevention
Keywords: Pre-Exposure Prophylaxis (PrEP); Antiretroviral therapy; Tenofovir Disoproxil Fumarate/Lamivudine/Dolutegravir
MeSH Terms: interventions — Lamivudine; dolutegravir

STUDY DESIGN:
Intervention Model Description: Oral - 1 tablet (300/300/50 mg TDF/3TC/DTG) daily
Masking Description: Age ≥ 15 years, inclusive, at the time of signing the informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TLD - Tenofovir Disoproxil Fumarate / Lamivudine / Dolutegravir (Experimental): The IMP is defined as any investigational marketed product to be administered to a study participant according to the study protocol.
  Participants will all receive TLD as detailed below. Treatment will be open-label, and drugs will be dispensed at intervals as specified in the Schedule of Events.
  Investigational Product Tenofovir disoproxil fumarate / lamivudine / dolutegravir Dosage Formulation 300 mg / 300 mg / 50 mg fixed dose combination tablet Route of Administration Oral Dosing Instructions 1 tablet (300/300/50 mg TDF/3TC/DTG) daily
  Interventions: Drug: TLD - Tenofovir Disoproxil Fumarate / Lamivudine / Dolutegravir

INTERVENTIONS:
Drug: TLD - Tenofovir Disoproxil Fumarate / Lamivudine / Dolutegravir — Dolutegravir, lamivudine and tenofovir disoproxil fumarate tablets, a combination of dolutegravir (integrase strand transfer inhibitor [INSTI]), lamivudine, and tenofovir disoproxil fumarate (both nucleoside reverse transcriptase inhibitors), is indicated as a complete regimen for the treatment of HIV-1 infection in adults and pediatric patients weighing at least 35 kg
  Other Names: Acriptega

SUMMARY:
This is a single-arm, open-label, effectiveness study designed to evaluate the use of Tenofovir, Lamivudine, and Dolutegravir in people with newly diagnosed HIV-1 infection initiating first-line Antiretroviral Therapy with Cabotegravir-Long-acting Pre-Exposure Prophylaxis exposure in the preceding 12 months. Participants will be followed up for a period of 12 months from enrolment.

DETAILED DESCRIPTION:
Study participants are HIV-1 infected adult patients recruited. A target of 100 participants will be enrolled and started on Tenofovir, Lamivudine, and Dolutegravir at enrolment. Clinical assessments for these participants will be conducted throughout the study as per the Schedule of Events.

This will be a two-phase interventional study to identify the optimally safe and effective Antiretroviral Therapy regimen for individuals with newly detected Human Immunodeficiency Virus infection after Cabotegravir-Long-acting Pre-Exposure Prophylaxis exposure. In the Initial Phase, the investigator will demonstrate proof of principle for the use of standardized Antiretroviral Therapy regimens in combination with pre-treatment genotypic drug resistance testing to achieve virologic suppression in individuals with prior Cabotegravir-Long-acting Pre-Exposure Prophylaxis exposure and understand drug resistance patterns prior to Antiretroviral Therapy initiation. To do this, the investigator will use a single-arm, interventional design using Tenofovir, Lamivudine, and dolutegravir. This supports programmatic rollout, particularly in developing countries where baseline Human Immunodeficiency Virus genotyping is not performed prior to initiation of Antiretroviral Therapy. The over-arching goals of Phase I are to determine the feasibility of our study design to recruit people with detectable Human Immunodeficiency Virus after prior use of Cabotegravir-Long-acting Pre-Exposure Prophylaxis failure and to estimate virologic suppression rates with current first-line standard of care, Tenofovir, Lamivudine, and Dolutegravir therapy.

At the conclusion of the Initial Phase, data will be assessed to determine the need for and optimal design of a potential Second Phase (the details of which will not be described in this protocol). Should the investigator find sub-optimal virologic suppression rates on Tenofovir, Lamivudine, and Dolutegravir regimens in this trial, the investigator would then proceed to the Second Phase in which the investigator will compare Darunavir/Ritonavir based Antiretroviral Therapy with Tenofovir, Lamivudine, and Dolutegravir in an open-label randomized, non-inferiority clinical trial. The aim of the second phase will be to determine whether an alternative to the predominant first-line regimen in much of the world will be required to optimise virologic suppression for this population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Age ≥ 15 years, inclusive, at the time of signing the informed consent.
3. Body weight ≥ 35 kg.
4. Confirmed HIV-1 infection.
5. Exposure to at least one dose of CAB-LA PrEP in the past 12 months.
6. Consent to initiation of ART.
7. Estimated glomerular filtration rate (eGFR) > 50 min/mL

Exclusion Criteria:

1. Any previous exposure to DTG.
2. Concurrent or recent (within the preceding 3 months) participation in another interventional clinical trial with a compound likely to interfere with any of the investigational medicinal products.
3. Known hypersensitivity or specific contraindications to the use of any of the active drugs in the treatment arms or similar compounds.
4. Is receiving or has received the following agents within 28 days prior to screening, and cannot discontinue their use for the duration of the study:

   1. tuberculosis therapy (i.e., rifampicin, rifapentine, rifabutin), with the exception of isoniazid (INH) prevention therapy;
   2. anti-convulsants (e.g., carbamazepine, oxcarbazepine, phenobarbital, phenytoin);
   3. herbal products (e.g., St John's Wort).
5. Any surgical or medical condition which may significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the safety of the volunteer or the objectives of the study or impair their ability to comply with the dosing schedule and/or protocol evaluations. The Investigator should make this determination in consideration of the volunteer's medical history.
6. Participant is judged by the Investigator to be at significant risk of failing to comply with the provisions of the protocol as to cause harm to self or seriously interfere with the validity of the study results. This including inability or an unwillingness to be followed up for the study period.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of TLD as first-line antiretroviral therapy (ART) in participants with HIV-1 infection and CAB-LA PrEP exposure in the past 12 months | At 6 Months
  Proportion of participants with virologic suppression (plasma HIV-1 RNA levels < 50 cp/mL) at Month 6

SECONDARY OUTCOMES:
To describe the epidemiology (i.e., prevalence and correlates) of HIV drug resistance patterns in participants with HIV-1 infection and prior CAB-LA PrEP exposure | 6 and 12 Months
  Proportion of participants with unsuppressed viral loads (HIV-1 RNA levels ≥ 50 cp/mL and ≥ 1000 cp/mL) at Month 6 and Month 12
To describe the epidemiology (i.e., prevalence and correlates) of HIV drug resistance patterns in participants with HIV-1 infection and prior CAB-LA PrEP exposure | 12 Months
  Time to virologic suppression
To describe the epidemiology (i.e., prevalence and correlates) of HIV drug resistance patterns in participants with HIV-1 infection and prior CAB-LA PrEP exposure | 12 Months
  Prevalence of HIV genotypic resistance to NRTI and INSTI drug classes at screening (baseline)
To describe the epidemiology (i.e., prevalence and correlates) of HIV drug resistance patterns in participants with HIV-1 infection and prior CAB-LA PrEP exposure | 12 Months
  Comparative prevalence of INSTI drug resistance in those with HIV and CAB-LA exposure and HIV acquisition deemed to occur prior to initiation of PrEP, during PrEP therapy, or after cessation of therapy
To investigate the development of HIV drug resistance over the duration of the trial of HIV treatment with TLD | 12 Months
  Assessment of genotypic drug resistance in participants with confirmed virologic failure (HIV-1 RNA ≥ 200 cp/mL on 2 or more occasions) throughout study duration
To evaluate the safety of TLD over 12 months | 12 Months
  Incidence of SAEs and DAIDS-defined Grade 3 and Grade 4 AEs, throughout study duration, including AEs considered related to the IMP
To evaluate the safety of TLD over 12 months | 12 Months
  Proportion of participants discontinuing treatment due to AEs
To evaluate the safety of TLD over 12 months | 12 Months
  Assessment of absolute values and changes in laboratory parameters over 12 months

OTHER OUTCOMES:
To conduct investigation on the effects of IMP on metabolic health over 12 months | 12 Months
  Changes from baseline in BMI throughout the study
To conduct investigation on the effects of IMP on metabolic health over 12 months | 12 Months
  Changes from baseline in lipids throughout the study
To conduct investigation on the effects of IMP on metabolic health over 12 months | 12 Months
  Changes from baseline in HbA1C throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: FRANCOIS WD VENTER, PhD, Study Director — Ezintsha, a division of Wits Health Consortium
Locations (3):
- South Africa (3):
  - Ezintsha, a division of Wits Health Consortium, Johannesburg, Gauteng
  - Africa Health Research Institute (AHRI), Durban, KwaZulu-Natal
  - Desmond Tutu Health Foundation, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
The data that will be shared is all of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication
Access Criteria: Anyone who wishes to access the data